CLINICAL TRIAL: NCT06872398
Title: Medical Comorbidities in Bipolar Disorder : Clinical Validation of Risk Factors and Biomarkers to Improve Prevention and Treatment;
Brief Title: Medical Comorbidities in Bipolar Disorder
Acronym: BIPCOM
Status: Recruiting | Type: Observational
Sponsor: Fondation FondaMental (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-A02218-37
Record Dates: First submitted 2024-04-22; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Psychiatric Disorder
MeSH Terms: conditions — Mental Disorders | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The BIPCOM study will assess metabolic and inflammatory biomarkers in bipolar disorder. Core biomarkers include adiponectin/leptin ratio, ALT, AST, blood count, C-peptide, fasting glucose, GGT, HDL-cholesterol, hsCRP, oxidized LDL, and triglycerides. Additional biomarkers, such as albumin, cystatin-C, IL-6, IL-10, LDL-cholesterol, salivary cortisol, serum amyloid A, testosterone, thyroid antibodies, TNF-α, total cholesterol, TSH, uric acid, and ghrelin, will provide further insights into systemic inflammation, oxidative stress, lipid metabolism, and cardiovascular risk. This analysis aims to enhance understanding of metabolic comorbidities in bipolar disorder
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Bipolar patients: Individuals diagnosed with bipolar disorder type I (BP I), bipolar disorder type II (BP II), or bipolar disorder not otherwise specified (BP NOS). Eligible participants must be between 18 and 65 years old and have had at least one contact with a mental health service in the past year. All participants will be required to provide signed informed consent before inclusion.
  Exclusion criteria include severe psychiatric comorbidities such as schizophrenia spectrum disorders, severe cognitive impairment, or severe substance/alcohol abuse, assessed using specific scores on the AUDIT and DAST scales. Patients planning to relocate within the next year will also be excluded.
  Interventions: Other: Blood and saliva sampling

INTERVENTIONS:
Other: Blood and saliva sampling — Physical and biological evaluation at inclusion visit V0 and at follow up visit V1 (after 1 year).
  the biological evaluation includes blood and saliva sampling at the 2 visits.

SUMMARY:
Bipolar Disorder (BD) is a common, heritable, chronic, and recurrent disorder that represents a critical public health problem, due to its prevalence, its high degree of disability and psychiatric and MC (MC): these represent a significant additive burden for BD patients, with a large clinical heterogeneity and an urgent need for personalised treatment and management. BIPCOM overarching purpose is to study MC in people with BD and to improve diagnostic and treatment outcomes with a precision medicine approach targeting 3 objectives: (1) to identify prevalence rates, risk and protective factors and natural history of MC among subjects with BD, through analyses of the Nordic biobanks and medical registers Work Package WP(WP2) and a cross- sectional study exploiting existing datasets of patients with BD (WP3); (2) to conduct an Exploratory Clinical Study (ECS - WP4) involving 400 subjects (80 X 5 recruiting sites), to assess the overall clinical profile of these patients and quantify the 1-year incidence of specific risk factors for the onset of metabolic syndrome (MetS) (WP5); (3) to develop a Clinical Support Tool (CST), including a set of recommendations, to support individualized clinical decision-making in BD comorbidity management and improve prevention, early detection and effective treatment, while ensuring the translation of project results' into clinical practice (WP5 and 6). BIPCOM will be implemented through continuous consultations with stakeholders (scientific and patients' associations, users and families), for ensuring results' acceptability and transferability. The successful implementation of the project will have a significant impact upon the general health of people with BD, eventually leading to lower mortality rates and reduced incidence of severe disabilities, whilst providing reliable methods and tools for patients' stratification and personalized treatments.

DETAILED DESCRIPTION:
WP1: Project Management (Leader: P1-IT)

This WP ensures effective project coordination, quality control, and risk management. It includes:

* Organizing the Kick-off Meeting (KoM)
* Managing and monitoring project progress based on predefined indicators
* Developing a Data Management Plan (DMP) to define data collection, processing, sharing, and storage
* Addressing ethical issues to ensure compliance with regulations and obtaining necessary authorizations
* Overseeing risk assessment throughout the project
* Managing project reporting, including consortium agreements, ethical guidelines, and periodic reports

WP2: Training Set - Register Study (Leader: P3-SE) This WP leverages Swedish and Norwegian national health registries to analyze cases of bipolar disorder (BD) and its comorbidities, particularly metabolic syndrome (MetS).

* Identification of BD patients from national registries and analysis of co-existing medical conditions
* Development of machine learning (ML) models to predict MetS and related outcomes
* Application of ML models using Swedish and Norwegian datasets, validated with genetic data
* Outputs: Dataset linkage, reports on BD prevalence and comorbidities, risk stratification models, and open-access ML algorithms

WP3: Real-World Risk Factors Study (Leader: P2-DE) This WP gathers real-world clinical data from five European centers to analyze BD comorbidities.

* Creation of a database using electronic medical records from 1,500 BD patients
* Collection of 24 key socio-demographic and clinical variables, including medical history, psychiatric hospitalizations, metabolic indicators, and medication history
* Development of a real-world dataset to investigate changes in MetS risk factors in BD patients over time
* Outputs: Standardized data collection tools (Medical Record Abstraction Tool - MRAT), anonymized database, and analysis of risk factors

WP4: Exploratory Clinical Study (ECS) - Calibration Phase (Leader: P5-FR) This WP aims to validate data from WP2 and WP3 through a prospective clinical study conducted across five European sites.

* Preparatory phase: Development of protocols, recruitment procedures, and sample collection guidelines
* Patient recruitment and baseline assessments: 400 BD patients stratified by age, sex, and disease severity
* Cross-sectional assessment of MetS in BD patients, identifying common diagnostic patterns and risk factors
* One-year follow-up to monitor MetS progression and treatment impact
* Physical activity monitoring: Using digital tools (ActiGraph GT9X Link) to track sedentary behavior and its association with MetS
* Creation of the BIPCOM biobank, collecting biological samples for proteomics, metabolomics, and genetic analyses
* Outputs: Clinical dataset, biomarker reports, biobank setup, and final study analyses

WP5: Development and Validation of a Precision Medicine (PM) Tool (Leader: P4-NO) This WP focuses on developing predictive models and a Clinical Support Tool (CST) to enhance risk assessment and personalized care in BD patients with metabolic syndrome (MetS).

* Prediction Model Development (M13-36)

  o Creation of Polygenic Hazard Scores (PHS) to improve risk prediction beyond standard Polygenic Risk Scores (PRS).
  * Integration of genetic, clinical, and lifestyle data to develop machine learning (ML)-based multimodal stratification algorithms.
  * Model calibration using data from WP2, WP3, and WP4.
* Development of a Clinical Support Tool (CST) (M20-36)

  * A risk calculator for clinicians to assess comorbidity risk in BD.
  * CST components:

    1. Electronic risk assessment questionnaire for patients and clinicians.
    2. Best practice recommendations for managing comorbidities.
    3. Personalized educational materials outlining individual risk levels.
  * Refinement of the CST beta version with stakeholder input (WP6).
* Clinical Validation in Real-World Settings (M22-34)

  * Testing the CST in 5-10 patients per site from the WP4 Exploratory Clinical Study (ECS).
  * Retrospective validation of MetS prediction using ECS baseline data.
  * Prospective validation with clinicians assessing the tool's usability and impact.

WP6: Stakeholder Involvement and Participation (Leader: P1-IT) This WP ensures active involvement of patients, clinicians, and policymakers to optimize the implementation of PM approaches in BD care.

* Mobilization of an International Stakeholder Group (M1-36)

  * Establishment of a Patient and Caregiver Advisory Board (PCAB) to oversee recruitment, retention, and public engagement.
  * Creation of a Scientific Advisory Board (SAB) with leading BD experts.
  * Focus on patient empowerment and education for healthcare providers about PM in psychiatry.
* Focus Groups (M6-34)

  o Patient focus groups in five sites to assess perspectives on BD comorbidities, unmet needs, and care improvements.
  * Clinician focus groups to evaluate PM implementation in BD treatment.
  * Thematic analysis using nVIVO software, with data stored under GDPR compliance.
* CST Fine-Tuning (M32-36)

  * The CST (developed in WP5) will be refined based on stakeholder feedback.
  * The final version will include clinical decision-support recommendations to enhance BD comorbidity management.

WP7: Dissemination, Public Engagement, and Exploitation (Leader: P6-ES) This WP ensures effective knowledge transfer to the scientific community, policymakers, and the public.

* Dissemination and Public Engagement Planning (M1-2) o Strategy development for knowledge transfer across research, healthcare, and policy sectors.
* Website Development and Maintenance (M1-36)

  o Launch of a project website by M3 for real-time updates, publications, and events.
* Dissemination Activities (M1-36)

  * Scientific publications in top-tier and national journals.
  * Conference participation, including ICPerMed and BD-related congresses.
  * BIPCOM mid-term and final events in Frankfurt (M19) and Barcelona (M35).
* Public Engagement (M1-36)

  o Promotion via social media, press releases, and media outreach.
* Exploitation of Results (M12-M36) o Development of an exploitation plan for sustainable implementation of findings.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of BP I, BP II, or BP NOS
* Have had at least one contact with mental health services in the past year
* Be aged between 18 and 65 years old
* Have signed an informed consent

Exclusion Criteria:

* Projected move within the next year.
* Severe psychiatric comorbidities (schizophrenia spectrum disorders).
* Severe cognitive impairment.
* Severe substance or alcohol abuse: quantified by specific scores on the AUDIT and DAST.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: To ensure representation, BP patients will be stratified by age, sex, and disorder severity. Subjects will be divided into 8 groups, with 5 patients randomly selected from each group, totaling 20 men, 20 women, 20 subjects aged 18-45, 20 aged 46-65, 20 with severe BP, and 20 with non-severe BP.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-10-11 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Metabolic Syndrome (MetS) | 1 year follow-up
  Number of bipolar patients meeting MetS criteria (≥3 of 5 criteria)

SECONDARY OUTCOMES:
Risk Factors for Metabolic Syndrome | 1 year follow up
  Correlations between risk factors and MetS incidence
Evolution of Metabolic Syndrome | 1 year follow up
  Changes in MetS components from inclusion to follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Marion LEBOYER, MD PhD, Principal Investigator — Fondation FondaMental; Ophélia GODIN, PhD, Study Director — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- France, Créteil, France

IPD SHARING:
Plan to Share IPD: No